CLINICAL TRIAL: NCT02304913
Title: Hypoglossal Acupuncture for Dysgeusia in Gynecologic Cancer Patients Undergoing Chemotherapy: A Randomized Controlled Trial
Brief Title: Hypoglossal Acupuncture for Dysgeusia in Patients Undergoing Chemotherapy
Acronym: OralAcu
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Heidemarie Haller, Postdoctoral Research Fellow, Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14-5953-BO
Record Dates: First submitted 2014-11-19; First posted 2014-12-02 (Estimated); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Acupuncture; Taste Disorders; Dysgeusia; Chemotherapy; Cancer
MeSH Terms: conditions — Taste Disorders; Dysgeusia; Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Hypoglossal acupuncture (Experimental): Single treatment of hypoglossal needle acupuncture during the chemotherapy administration: Treated points will be Jinjin (Golden Liquid/EX-HN12) left beside the lingual frenulum and Yuye (Jade Fluid/EX-HN13) right beside the lingual frenulum. Both points are treated in quick succession with immediate removal of the needle.
  Interventions: Other: Hypoglossal acupuncture
- Sham acupuncture (Sham Comparator): Single treatment of hypoglossal sham acupuncture uring the chemotherapy administration: Treated points will be 1 to 1.5 cun (a cun is defined as the width of the patient's thumb at the knuckle) beside the verum acupuncture points Jinjin and Yuye using the dull side of the needle.
  Interventions: Other: Sham acupuncture
- Dietary recommendations (Active Comparator): This group adheres to specific dietary recommendations for dysgeusia of the German Cancer Society.
  Interventions: Behavioral: Dietary recommendations

INTERVENTIONS:
Other: Hypoglossal acupuncture
  Arms: Hypoglossal acupuncture
Other: Sham acupuncture
  Arms: Sham acupuncture
Behavioral: Dietary recommendations
  Arms: Dietary recommendations

SUMMARY:
This randomized controlled trial aims to investigate hypoglossal acupuncture in comparison to sham acupuncture and standard medical treatment (dietary recommendations) in the treatment of dysgeusia in cancer patients undergoing chemotherapy.

DETAILED DESCRIPTION:
Taste disorders are frequent side effects in patients undergoing chemotherapy (CTX). Dysguesia has prevalence rates of 16% to 1000% during CTX with sometimes also persistent courses. Impact of dysguesia on appetite, body weight as well as health-related quality of life was shown. Until now, evidence for adequate treatment options is limited to specific diary recommendations. Acupuncture in the treatment of side effects of chemotherapy was investigated for nausea and xerostomia, but not for dysguesia. Therefore, this randomized controlled trial aims to investigate hypoglossal acupuncture in comparison to sham acupuncture and standard medical treatment (dietary recommendations) in the treatment of dysgeusia in cancer patients undergoing chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Initial treatment with platinum-containing or taxane-based CTX (regardless of the the length of the CTX cycle)
* Senological, gynecological or internistic tumors
* Phantogeusia (on average ≥4 NRS)
* Willingness to participate in the study and written informed consent

Exclusion Criteria:

* Severe stomatitis
* Dysgeusia before the CTX based on neurological diseases, diabetes, or the ingestion of drugs with taste disorders as side effects
* Leucopenia/neutropenia
* Intake of anticoagulants
* Smoking
* Severe physical or mental comorbidity (due to which the patient is unable to participate in the study)
* Participation in other CAM treatments within the integrative oncology care
* Participation in other studies on the effectiveness of interventions for oral complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Dysgeusia (Phantogeusia) (NRS - Numeric Rating Scale) | 7 days

SECONDARY OUTCOMES:
Dysgeusia (Parageusia, Hypogeusia, Hypergeusia) (NRS - Numeric Rating Scale) | 7 days
Xerostomia (NRS - Numeric Rating Scale) | 7 days
Stomatitis (NRS - Numeric Rating Scale) | 7 days
Appetite (NRS - Numeric Rating Scale) | 7 days
Impairment (NRS - Numeric Rating Scale) | 7 days
Adverse Events (free text) | 7 days

OTHER OUTCOMES:
Treatment Expectancy and Credibility (TCS - Treatment Credibility Scale + BI - Blining Index) | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Gustav Dobos, Prof., MD, Study Director — Center for Integrative Medicine and Health, University Hospital Essen, University of Duisburg-Essen
Locations (3):
- Germany (3):
  - Department of Gynecology & Gynecologic Oncology, Evang. Kliniken Essen-Mitte, Essen, North Rhine-Westphalia
  - Universitätsklinikum Mannheim, Internistische Onkologie, Mannheim
  - Robert Bosch Krankenhaus Stuttgart, Stuttgart

REFERENCES:
- [Derived] Haller H, Wang T, Lauche R, Choi KE, Voiss P, Felber S, Cramer H, Ataseven B, Kummel S, Paul A, Dobos G. Hypoglossal acupuncture for acute chemotherapy-induced dysgeusia in patients with breast cancer: study protocol of a randomized, sham-controlled trial. Trials. 2019 Jul 4;20(1):398. doi: 10.1186/s13063-019-3525-y. PMID 31272494